CLINICAL TRIAL: NCT01921075
Title: Patterns and Plasticity of Orthotopic and Ectopic Fat Deposition and Associations With Insulin Sensitivity: A Magnetic-resonance-imaging and -Spectroscopy Study in Lean and Obese Individuals: Methodological Part
Brief Title: Physiologic Plasticity of Intramyocardial Lipid Storage
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 124/08; 1587 (Other: Inselspital)
Record Dates: First submitted 2013-08-05; First posted 2013-08-13 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Lipid Metabolism
Keywords: physiology, normal function
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Volunteers: young (age<30), healthy, lean (BMI<25) volunteers
  Interventions: Other: normal dietary behavior; Other: Magnetic resonance spectroscopy

INTERVENTIONS:
Other: normal dietary behavior — normal dietary behavior during examination days
Other: Magnetic resonance spectroscopy — Non-invasive diagnostic procedure

SUMMARY:
The main goal of the present study was to provide a technical basis for future studies assessing the role of cardiac lipids. More specifically, non-invasive MR-Spectroscopy (MRS) techniques will be used in this study to:

1. assess the methodological reproducibility of MRS-measurements of cardiac lipids in humans
2. investigate physiological variations of cardiac lipids by measuring day-to-day changes under identical conditions
3. determining diurnal variations of cardiac lipids in humans

DETAILED DESCRIPTION:
Background

Obesity is a well known risk factor for the development of glucose intolerance, type 2 diabetes mellitus and, consequently, diabetic complications like cardiovascular disease. Importantly, obesity is not only associated with lipid accumulation in adipose tissue (orthotopic fat deposition), but also in non-adipose tissues (ectopic fat deposition). Clinical studies have repetitively shown that muscular and hepatic lipid accumulation as well as elevated visceral adipose tissue is associated with the development of central and peripheral insulin resistance. In addition, recent data from animal studies show increasing evidence that two other organs, the heart and the pancreas, may also be involved in the pathophysiological processes of reduced insulin sensitivity. While reduced insulin secretion in the course of type 2 diabetes has been well documented, the importance of pancreatic fat deposition as an early step in this process has only recently been suggested based on animal models. Conversely, ischemic heart disease is one of the most dangerous complications of diabetes mellitus, its prevention thereby being a cornerstone of current diabetes management. Recent data suggest that changes in the lipid metabolism of the heart and associated epi- and myocardial lipid deposition may be earliest signs of diabetic cardiopathy.

Magnetic-Resonance-Imaging (MRI) and -Spectroscopy (MRS) are among the most versatile methods for non-invasive studies of human tissue and/or metabolism in vivo and in situ. The excellent soft tissue contrast of MRI has already led to the implementation of this method for the assessment of whole body lipid accumulation, whereas MRS has successfully been applied to study lipid metabolism of skeletal muscle and liver. The extended application of this method towards heart and pancreas will allow a comprehensive investigation of orthotopic and ectopic fat deposition in humans and its association with the development of insulin resistance and diabetes mellitus.

The methodological part of the study will focus on the physiologic plasticity of cardiac lipids in order to assess:

i) methodological reproducibility ii) intra-individual physiological reproducibility by measuring day-to-day variations as well as variations during the day.

Objective

i) Adapting and optimizing the single-voxel MRS sequence that is currently used for muscle and liver, such that respiratory and cardiac double-triggering enables spectroscopy of the cardiac muscle.

ii) Validate the methodology under different standardized physiologic conditions.

Methods

Cardiac lipids are determined during five independent MR-examinations distributed over two days separated by one or two weeks. Both days included a measurement in the morning after an overnight fast (>8h) and one in the afternoon (8h after breakfast, 3.5h after lunch). To determine methodological reproducibility, the afternoon measurement was repeated on one of the two days (1h break). Preparation of the volunteers included perpetuation of their normal diet, but restricted physical activity for two preceding days. Cardiac lipids were determined by single-voxel MR-Spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* male
* age 18-30
* BMI <25
* healthy
* written informed consent

Exclusion Criteria:

* contraindications to MRI examinations (claustrophobia, implanted devices (pacemaker, insulin pump, neurostimulators))

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: males between the age of 18 and 30 years with either a BMI of 18-24
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Intramyocardial lipid content | at baseline (morning of examination day 1)

SECONDARY OUTCOMES:
Intramyocardial lipid content | evening of examination day 1, i.e. 8 hours after baseline
Intramyocardial lipid content | morning of examination day 2, i.e. 7 days after baseline
Intramyocardial lipid content | evening of examination day 2, i.e. 7 days & 8 hours after baseline
Intra-individual variation of intramyocardial lipid content | evening of examination day one, i.e. 8 hours after baseline
  Difference between evening and morning measurement within examination day one
Intra-individual variation of intramyocardial lipid content | evening of examination day two, i.e. 7 days & 8 hours after baseline
  Difference between evening and morning measurement within examination day two
Intra-individual difference of intramyocardial lipid content (morning) over one week | morning of examination day one, i.e. 7 days after baseline
  Difference between morning measurements of examination day 1 and examination day 2

CONTACTS AND LOCATIONS:
Overall Officials: Ith, PhD & MD/PhD, Principal Investigator — University Institute of Diagnostic Interventional and Pediatric Radiology of the Inselspital Bern
Locations (1):
- Institute of Diagnostic Interventional and Pediatric Radiology, University Hospital Bern, Bern, Switzerland